CLINICAL TRIAL: NCT00895700
Title: WEB-based Distress Management Program for Implantable CARdioverter dEfibrillator Patients (WEBCARE) Trial
Brief Title: Internet-based Intervention in Cardioverter-defibrillator Patients to Enhance Quality of Life
Acronym: WEBCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tilburg University (Other)
Collaborators: Erasmus Medical Center (Other); Amphia Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Canisius-Wilhelmina Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Vlietland Ziekenhuis (Other)
Responsible Party: Principal Investigator, Dr. SS Pedersen, Professor of cardiac psychology, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UVT-MP-001
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Heart Diseases; Implantable Cardioverter-Defibrillators
Keywords: Anxiety; ICD concerns; Quality of life
MeSH Terms: conditions — Heart Diseases; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based behavioral intervention (Experimental)
  Interventions: Behavioral: web-based multifactorial intervention
- Usual care (No Intervention)
  Interventions: Behavioral: web-based multifactorial intervention

INTERVENTIONS:
Behavioral: web-based multifactorial intervention — 12-week multi-factorial web-based behavioral intervention comprised of psycho-education, cognitive behavioral therapy (CBT) and relaxation therapy
  Other Names: Psycho-education; Cognitive behavioral therapy; Relaxation therapy

SUMMARY:
The implantable cardioverter defibrillator (ICD) is generally well-accepted by patients, but a subgroup experiences increased anxiety and poor quality of life. A web-based behavioral intervention may comprise a novel approach to reduce anxiety and enhance well-being in ICD patients, which may be equally effective and have advantages over more traditional forms of therapy, due to its low-threshold accessibility via the internet.

The purpose of this study is to determine whether patients receiving a behavioral intervention via the internet experience less anxiety and device concerns and improved quality of life compared to patients receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* patients implanted with a cardioverter-defibrillator (ICD)
* between 18-75 years of age
* speaking and understanding Dutch
* with access to the internet and ability to use the internet
* providing written informed consent

Exclusion Criteria:

* a life expectancy less than 1 year
* a history of psychiatric illness other than affective/anxiety disorders
* on the waiting list for heart transplantation
* with insufficient knowledge of the Dutch language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline
Anxiety | 14 weeks
Anxiet | 26 weeks
Anxiety | 52 weeks

SECONDARY OUTCOMES:
Cortisol awakening response | Baseline
Cortisol awakening response | 14 weeks
Cortisol awakening response | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susanne S Pedersen, PhD, Principal Investigator — Tilburg University, The Netherlands
Locations (6):
- Netherlands (6):
  - Canisius-Wilhelmina Hospital, Nijmegen, Gelderland
  - Amphia Hospital, Breda, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Vlietland Ziekenhuis, Schiedam

REFERENCES:
- [Derived] Habibovic M, Broers E, Heumen D, Widdershoven J, Pedersen SS, Denollet J. Optimism as predictor of patient-reported outcomes in patients with an implantable cardioverter defibrillator (data from the WEBCARE study). Gen Hosp Psychiatry. 2018 Jan-Feb;50:90-95. doi: 10.1016/j.genhosppsych.2017.10.005. Epub 2017 Nov 8. PMID 29127812
- [Derived] Habibovic M, Denollet J, Cuijpers P, van der Voort PH, Herrman JP, Bouwels L, Valk SD, Alings M, Theuns DA, Pedersen SS. Web-based distress management for implantable cardioverter defibrillator patients: A randomized controlled trial. Health Psychol. 2017 Apr;36(4):392-401. doi: 10.1037/hea0000451. Epub 2017 Feb 13. PMID 28192003
- [Derived] Habibovic M, Denollet J, Cuijpers P, Spek VR, van den Broek KC, Warmerdam L, van der Voort PH, Herrman JP, Bouwels L, Valk SS, Alings M, Theuns DA, Pedersen SS. E-health to manage distress in patients with an implantable cardioverter-defibrillator: primary results of the WEBCARE trial. Psychosom Med. 2014 Oct;76(8):593-602. doi: 10.1097/PSY.0000000000000096. PMID 25264974
- [Derived] Habibovic M, Cuijpers P, Alings M, van der Voort P, Theuns D, Bouwels L, Herrman JP, Valk S, Pedersen S. Attrition and adherence in a WEB-Based Distress Management Program for Implantable Cardioverter defibrillator Patients (WEBCARE): randomized controlled trial. J Med Internet Res. 2014 Feb 28;16(2):e52. doi: 10.2196/jmir.2809. PMID 24583632
- [Derived] Pedersen SS, Spek V, Theuns DA, Alings M, van der Voort P, Jordaens L, Cuijpers P, Denollet J, van den Broek KC. Rationale and design of WEBCARE: a randomized, controlled, web-based behavioral intervention trial in cardioverter-defibrillator patients to reduce anxiety and device concerns and enhance quality of life. Trials. 2009 Dec 23;10:120. doi: 10.1186/1745-6215-10-120. PMID 20030843